CLINICAL TRIAL: NCT04111913
Title: An Open, Single-arm, Multi-center Exploratory Study of Sequential Anlotinib Followed by EP Regimen Plus Concurrent Radiotherapy for Unresectable Stage III Non-small Cell Lung Cancer
Brief Title: A Study of Sequential Anlotinib Followed by EP Regimen Plus Concurrent Radiotherapy for Unresectable Stage III Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L028
Record Dates: First submitted 2019-09-25; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-08

CONDITIONS: Unresectable Stage III Non-small Cell Lung Cancer
Keywords: anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib and chemoradiotherapy (Experimental): anlotinib: 12 mg, po, qd, on day1-14 of a 21 days cycle; anlotinib will be administrated to 2 cycles for induction before the 2 cycles of chemoradiation and anlotinib will be administrated up to 1year or disease progression for maintenance treatment.
  EP regimen: cisplatin 50mg/m2, d1, 8, 29, 36; etoposide 50mg/m2, d1~5, d29~33. Radiotherapy program: 2 Gy / time / d, 5 d / week;PTV radiotherapy 60~66Gy/30~33 times/6~7 weeks.
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — anlotinib once daily on days 1-14 of 21days cycle.

SUMMARY:
Anlotibib (AL3818) is a kind of innovative medicines approved by State Food and Drug Administration（SFDA:2011L00661） which was researched by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd. Anlotinib is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR2、VEGFR3、PDGFRβ and c-Kit. It has the obvious resistance to new angiogenesis. The trial is to evaluate the efficacy and safety of sequential anlotinib followed by EP regimen plus concurrent radiotherapy for unresectable stage III non-small cell lung cancer(NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure.
2. ≥ 18 and ≤ 70 years of age within male and female.
3. Histologically confirmed，locally advanced NSCLC of stage IIIA/IIIB.
4. Unresectable stage IIIA and stage IIIB with pathological evidence of the following images or lymph nodes:

   1. Multiple metastases of the mediastinal lymph nodes are transferred into a massive mass or multiple sites (IIIA: T1-3N2 or IIIB: T4N2)
   2. Contralateral hilar, mediastinal lymph nodes, or the same, contralateral scalene or supraclavicular lymph node metastasis (IIIB: T1-4N3)
   3. The lesion invades the heart, aorta and esophagus (IIIB: T4N0-1)
5. Life expectancy of more than 3 months.
6. Eastern Cooperative Oncology Group(ECOG)performance scale 0-1.
7. Weight loss ≤5% in the last 3 months since enrollment.
8. Good lung function (predicted FEV1 ≥1 liter), no history of bronchial pneumonia, tracheobronchial disease and upper respiratory tract bleeding.
9. None previous chemotherapy or targeted therapy.
10. Adequate hepatic, renal, heart, and hematologic functions (Absolute Neutrophil Count(ANC) ≥ 1.5×109/L, Platelet (PLT) ≥ 100×109/L, Hemoglobin(HB) ≥ 90 g/L, total bilirubin within 1.5×the upper limit of normal(ULN), and serum transaminase≤2.5×the Upper Limit Of Normal(ULN), serum creatine ≤ 1.25 x Upper Limit Of Normal(ULN), creatinine clearance rate ≥ 45ml/min.
11. For women of child-bearing age, the pregnancy test results (serum or urine) within 7 days before enrolment must be negative. They will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men (previous surgical sterilization accepted), will take appropriate methods for contraception during the study until the 8th week post the last administration of study drug.

Exclusion Criteria:

1. small cell lung cancer (including small cell and non-small cell mixed lung cancer).
2. Radiologically documented evidence of tumor lesions from large vessels ≤ 5mm or major blood vessel invasion or encasement by cancer; Obvious cavity or necrosis formed in the tumor.
3. History and complication:

   1. Less than 4 weeks from the last clinical trial or participating in other clinical studies.
   2. Other active malignancies that require simultaneous treatment.
   3. History of malignancy except cured basal cell skin cancer, or carcinoma in situ of the cervix, or superficial bladder cancer.
   4. Patients with previous anti-tumor treatment-related adverse reactions (excluding hair loss) did not return to NCI-CTCAE ≤ 1 level.
   5. Coagulation disfunction（INR>1.5 or PT>Upper Limit Of Normal(ULN)+4s or Activated Partial Thromboplastin Time (APTT) >1.5 Upper Limit Of Normal(ULN)）, hemorrhagic tendency or receiving the therapy of thrombolysis or anticoagulation.
   6. Renal insufficiency. Urine protein≥++, and 24h urine protein quantitation≥1.0g.
   7. Patients had major surgery or severe trauma before enrollment. The effects of surgery or trauma have been eliminated for less than 14 days.
   8. Severe acute or chronic infection requiring systemic treatment.
   9. Patients who suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female ≥ 470 ms). Grade III-IV cardiac insufficiency according to New York Heart Association(NYHA) criteria or echocardiography check: left ventricular ejection fraction (LVEF)<50%.
   10. Peripheral neuropathy with ≥CTCAE 2 degrees currently present, except for trauma.
   11. Respiratory syndrome (≥CTC AE grade 2 dyspnea).
   12. Symptomatic serous effusion requiring treatment .(including hydrothorax, ascites, hydropericardium)
   13. Long-term untreated wounds or fractures（in addition to tumor-induced pathological fractures).
   14. Decompensated diabetes or other remedies for high-dose glucocorticoid therapy.
   15. Significant factors that influence the ingestion and absorption of medicine, (e.g. unable swallow, chronic diarrhea and intestinal obstruction.
   16. Clinically significant hemoptysis occurred within 3 months prior to enrollment (daily hemoptysis greater than 50 ml). History of clinically relevant major bleeding event=<3 months (e.g. gastrointestinal hemorrhage, Hemorrhagic acne， bleeding gastric ulcer, occult blood test ≥ (++), and vasculitis.
   17. Planned systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, immunotherapy, within 4 weeks prior to enrollment in other anti-cancer drug clinical trials or within 4 weeks prior to grouping or during the study.
4. Physical examination and laboratory inspection:

   1. Have a positive history of human immunodeficiency virus (HIV) test or have acquired immunodeficiency syndrome (AIDS).
   2. Untreated active hepatitis (Hepatitis B: HBsAg-positive and HBV DNA ≥ 500IU/mL; Hepatitis C: HCV RNA-positive and abnormal liver function); Combined hepatitis B and C infection
5. At the discretion of the investigator, the patient may have other factors that may cause the study to be terminated midway, such as other serious illnesses or serious laboratory abnormalities or other safety that may affect the subject, or test data and samples. Factors such as family or society collected.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival (PFS) | Approximately 12 months.
  Progression-Free Survival (PFS) as Assessed by Investigator Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1)

SECONDARY OUTCOMES:
The recurrence rate in 12-month | 12 months.
  The proportion of patients with disease progression within 12 months of the initiation of consolidation treatment with anlotinib.
The recurrence rate in 24-month | 12 months.
  The proportion of patients with disease progression within 24 months of the initiation of consolidation treatment with anlotinib.
The disease control rate in 6-month | 6 months.
  The proportion of CR, PR, and SD within 6 months of the initiation of consolidation treatment with anlotinib.
The disease control rate in 12-month | 12 months.
  The proportion of CR, PR, and SD within 12 months of the initiation of consolidation treatment with anlotinib.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China